CLINICAL TRIAL: NCT00659321
Title: Placebokontrollierte Untersuchung Zur Wirkung Von Nikotinsäure Auf Die Dyslipidämie Bei Metabolischem Syndrom Und Das Arterioskleroserisiko (Placebo Controlled Investigation of Efficacy of Nicotine Acid on Dyslipidaemia in Patients With Metabolic Syndrome and the Risk of Atherosclerosis)
Brief Title: Efficacy of Nicotine Acid on Dyslipidaemia in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Technische Universität Dresden (Other); University of Regensburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIASPAN-DD-2005
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Metabolic Syndrome; Dyslipidaemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): 16 weeks, randomisation with 500 mg, after 4 weeks elevation of 1000 mg, after week 8 to week 16 1500 mg study medication
  Interventions: Drug: nicotine acid
- 2 (Placebo Comparator): 16 weeks treatment with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nicotine acid — 16 weeks, randomisation with 500 mg, after 4 weeks elevation of 1000 mg, after week 8 to week 16 1500 mg study medication
  Arms: 1
Drug: placebo — 16 weeks treatment with placebo
  Arms: 2

SUMMARY:
Placebo controlled evaluation of effectiveness of nicotine acid in treatment of postprandial dyslipidemia in patients with metabolic syndrome. Nicotine acid decreases postprandial hyperlipidaemia in patients with metabolic syndrome which reduces the low-grade inflammation and the risk of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* dyslipidemia (triglycerides >= 150 mg/dl and/or decreased levels of HDL-cholesterol <40 mg/dl in men or < 50 mg/dl in women)
* further components of the metabolic syndrome: Hypertension: blood pressure >= 130/85 mmHg or/and Hyperglycemia: fasting plasma glucose >= 100 mg/dl or/and 2 hour plasma glucose after 75g glucose load (OGTT) >= 140 mg/dl or/and Obesity: waist circumferences > 102 cm in men or >88 cm in women

Exclusion Criteria:

* Contraindication and incompatibility of nicotine acid
* Patients with ulcus ventriculi or ulcus duodeni
* Intake of lipid lowering drugs < 6 weeks before randomization
* therapy of type 2 diabetes with insulin, glitazones, acarbose or more than one antidiabetic drug (only mono-therapy with metformin or sulfonyl urea is permit) - no acceptable therapy of diabetes with levels of HbA1C>=8.0%
* cardiovascular events in the last 6 months
* chronic inflammatory diseases (lupus erythematodes, arthritis, morbus Crohn or colitis ulcerosa)
* ALAT elevation 2.5 times more than the normal limit
* pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Placebo controlled evaluation of effectiveness of nicotine acid in treatment of postprandial dyslipidemia in patients with metabolic syndrome | after 16 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Markolf Hanefeld, MD, PhD, Principal Investigator — GWT-TUD GmbH
Locations (1):
- GWT-TUD GmbH, Centre for Clinical Studies, Dresden, Germany